CLINICAL TRIAL: NCT07116746
Title: A Phase 2, Multicenter, Open-label, Efficacy and Safety Study of AR882 and XOI Co-administration in Participants With Uncontrolled Gout Who Have Previously Failed Uricase Treatment
Brief Title: Evaluation of Efficacy and Safety of AR882 and XOI Co-administration in Uricase Treatment Failed Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Arthrosi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AR882-204
Record Dates: First submitted 2025-08-07; First posted 2025-08-12 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Gout; Gouty Arthritis; Hyperuricemia; Gout Chronic; Refractory Gout; Uncontrolled Gout; Tophaceous Gout
Keywords: Uricase Failure; Pegloticase Failure; Krystexxa Failure; Rasburicase Failure
MeSH Terms: conditions — Gout; Arthritis, Gouty; Hyperuricemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AR882 75 mg + XOI (Experimental): AR882 75 mg plus XOI low dose taken once daily starting on Day 1 for 2 weeks then titrate up to AR882 75 mg plus XOI high dose taken once daily for duration of 6-month treatment period in the Core Study Phase. Participants who complete the Core Study Phase can opt in to the Optional Extension Phase and continue to receive AR882 75 mg plus XOI high dose taken once daily for duration of an additional 6-month treatment period.
  Interventions: Drug: AR882 75 mg; Drug: XOI Low Dose; Drug: XOI High Dose

INTERVENTIONS:
Drug: AR882 75 mg — Solid Oral Capsule
Drug: XOI Low Dose — Solid Oral Tablet
Drug: XOI High Dose — Solid Oral Tablet

SUMMARY:
This study will assess the effect of AR882 and XOI co-administration on sUA lowering as well as reducing tophus burden in the population that has failed uricase treatment (eg., pegloticase). Failed uricase treatment is defined as having an inherent intolerance, anaphylaxis, infusion reaction, antibody development, and/or at least one sUA level that rose to greater than 6 mg/dL while on therapy.

ELIGIBILITY:
Inclusion Criteria:

* History of uncontrolled gout
* Presence of ≥1 clinically visible tophus
* Last uricase infusion occurred ≥3 months
* Body weight no less than 50 kg
* Serum creatinine must be < 3.0 mg/dL and estimated CLcr ≥ 40 mL/min

Exclusion Criteria:

* Malignancy within 5 years, except for successfully treated basal or squamous cell carcinoma of the skin
* Pregnant or breastfeeding
* History of symptomatic kidney stones within the past 6 months
* Received pegloticase, rasburicase or other experimental uricases within the last 3 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Serum urate (uric acid) (sUA) level < 6 mg/dL at month 6 | 24 weeks
  Proportion of patients with serum urate (uric acid) (sUA) level < 6 mg/dL at month 6

SECONDARY OUTCOMES:
Change in tophus burden by month 6 | 24 weeks
  Change in tophus burden by measurement of targeted tophi area at Month 6
Incidence of Adverse Events | 56 weeks
  Treatment Emergent Adverse Events and Serious Adverse Event incidence

CONTACTS AND LOCATIONS:
Overall Officials: Robert Keenan, MD, Study Director — Arthrosi Therapeutics, Inc.
Locations (4):
- United States (4):
  - Arthrosi Investigative Site (105), Margate, Florida
  - Arthrosi Investigative Site (102), Miami, Florida
  - Arthrosi Investigative Site (103), Duncansville, Pennsylvania
  - Arthrosi Investigative Site (104), West Lake Hills, Texas

IPD SHARING:
Plan to Share IPD: No